CLINICAL TRIAL: NCT04399616
Title: Map of Risks in Home Care From Primary Health Care.
Brief Title: Map of Risks in Home Care From Primary Health Care, an Approach From Health Care Quality.
Acronym: ATDOM_SP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R19/006
Record Dates: First submitted 2020-03-24; First posted 2020-05-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-02

CONDITIONS: Community Health Services
Keywords: Patient Safety; Quality of Healthcare; Information Technology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The intervention consists of the availability in the patient's medical history of the visual risk map. The patients in the intervention group will have a risk map in their medical history similar to the one presented in image (annex 2), and any care provider will have immediate access to this map which we think will help them to prioritize the implementation of the relevant practices. safe (in relation to the areas that appear in red).
  Areas of risk:
  Other independent variables will be the areas of risk:
  * Identification of the patient
  * Functional autonomy and quality of life
  * Caregiver
  * Safe management and use of medicines
  * Risk of falls
  * Risk of injuries and pressure ulcers
  * Symptom control
  * Risk of infection associated with health care
  * Patient and family values and beliefs
  * Social risk
  * Unplanned hospital admissions / proactive monitoring
  * Continuity of care 7X24 h
  * Transfers (between care levels)
  * Safety culture
  * Nursing work environment
  Interventions: Other: Risk Map
- No intervention (No Intervention): The patients in the control group will have in their medical records the usual records of the comprehensive geriatric assessment.

INTERVENTIONS:
Other: Risk Map — The tool we test in this project (the visual hazard map) aims to enable the practitioner to quickly identify critical areas for systematically implementing relevant safe practices (appropriate for each situation).
  Arms: Experimental

SUMMARY:
Background: Home health care is very complex. The registration of many disassembled information makes it difficult to interpret and does not allow the identification of critical areas for risk management.

Hypothesis / Research question: The availability of a risk map, with visual alerts to identify the critical areas, will facilitate the implementation of safe practices and improve the safety of patients included in the DOMicillary care program (ATDOM).

Objectives: To design and evaluate the effectiveness of the availability of a Visual Risks Map (MRV) in the computerized medical histories of ATDOM patients in the improvement of their safety and quality of life.(QL).

Methods: Once MRV is designed, the investigators will conduct a randomized clinical trial by conglomerates (Primary Care centers) to evaluate whether the fact of having this MRV (intervention) in the medical histories of ATDOM patients reduces avoidable income, falls and wounds and improves QL.

Analysis plan: Baseline description: socio-demographic characteristics, risk's levels in the different areas and other covariates in the control and intervention groups. Chi-square test to compare frequency of outcomes between control and intervention groups. Cox regression model to estimate time until the outcomes appear, adjusting for the different variables.

Expected results: The frequency of avoidable hospital admissions / emergencies' visits, falls and sores / infections will be significantly lower in the group of patients who have MRV in their clinical histories. Their qL wil be better.

Applicability and Relevance: It is a feasible and easy-to-implement project. It provides a practical utility for a lot of information that the investigators record and affects a key aspect of quality of care.

DETAILED DESCRIPTION:
Design:1st phase: Visual Risk Map Design (MRV); 2nd Phase: Randomized clinical trial by conglomerates (Primary Care Centers).

Study population (indicate inclusion and exclusion criteria):

Patients included in the Home Care program (ATDOM) assigned to the Primary Care Centers in the territory who agree to participate in the study. The only exclusion criterion will be the patient's refusal to participate in the study

Sample size and sampling procedure:

The study will be conducted in 8 Centers; 4 will be randomly assigned to intervention and 4 to control. If approximately 80% of patients have had an admission in the previous year and the investigators intend that, with our intervention, this percentage drops to 70%, for a confidence of 95% (alpha error of 5%) and a statistical power of 80%, the investigators will need a sample of 231 patients and, if the investigators have a 15% loss, 272 patients per group (control and intervention). Each Center will be able to provide approximately 50 ATDOM patients. All patients will be invited to participate. They will be given a brief explanation of the study and invited to sign informed consent (in case the patient has a significant cognitive impairment, their guardian will sign the consent). All patients who meet inclusion criteria will be included.The basic morbidity and mortality characteristics of the sample will be compared with the MSIQ (health and quality monitoring) record of CatSalut (catalonia health services).

Dependent and independent variables (for quantitative studies):

Dependent variables: Percentage of patients with: hospital admissions / avoidable hospital emergency room visits (main variable) during the follow-up year sores falls. Death and final institutionalization will also be considered dependent variables In addition to the percentage of patients with admissions, the investigators will also consider the total number of preventable admissions and visits to hospital emergencies during the follow-up period. Another dependent variable will be the quality of life, which the investigators will measure using the EuroQol-5D index (see appendix 1), a record currently available at the e-cap clinical station.

Independent variables: The main independent variable is "intervention".

Intervention: The intervention consists of the availability in the patient's medical history of the visual risk map. Patients in the intervention group will have a risk map in their medical history and any professional who treats them will have immediate access to this map, which the investigators think will help them prioritize the implementation of the relevant practices. safe (in relation to the areas that appear in red) Patients in the control group will have in their clinical histories the usual records of comprehensive geriatric assessment

Risk areas: Other independent variables will be the risk areas: Patient identification, Functional autonomy and quality of life, Caregiver, Management and safe use of medications, Risk of falls, Risk of pressure injuries and ulcers, Control of symptoms, Risk of infection associated with health care, Values and beliefs of the patient and the family, Social risk, Unplanned hospital admissions / proactive follow-up, Continuity of care 7 days X 24 hours , Transfers (between levels of care), Security culture and Nursing work environment.

During the first stage of the project, the 15 variables (indicators) corresponding to the aforementioned Risk Areas (RAs) will be created based on the integration of one or more variables. the investigators detail all the "primary" variables that will be considered for inclusion in the 15 indicators ("secondary" variables) corresponding to the 15 RAs, which will generate 1 synthetic indicator of the overall risk of the patient. The selection of the variables to be included was made based on the bibliographic search; their final inclusion and the relative contribution of each will depend on the consensus among the members of the interdisciplinary team of professionals (doctors, nurses, social workers) experts in ATDOM. For the weighting (contribution of each of the variables to the final indicator) will be taken into account on the one hand the magnitude / severity of the problem measured by the variable and on the other the existence of feasible interventions (safe practices) that have proven its effectiveness in improving it. The same team will also decide the cut points; that is, from which values of the new variables / indicators (operated from the weighted "primary" variables) is it considered moderate risk and when it goes to high risk. For this recoding and fusion of primary variables will have the support of a mathematical expert and the professionals of the Technologies of the Information and the Communication (TIC) will be the commissions.

Most of the data will be collected from the records in the e-cap (primary care clinical station): socio-demographic variables, scores at different scales, diagnostic codes. Other sources of information will be direct observation, interviews with patients and caregivers, exchange of information with other professionals involved (social services, professionals from other care devices ...).

Once the first phase of the study has been completed with the "construction" of the 15 variables corresponding to the risk areas, the investigators will make a descriptive analysis: the investigators will determine the mean and standard deviation for quantitative variables and frequencies (percentages) for qualitative ones. Based on the categorization of risk areas, the investigators will analyze the distribution of these categories (low, moderate or high risk) for each of the 15 RAs.

The investigators will do a baseline comparative analysis (using Chi-square test and Student's t, as the investigators compare qualitative or quantitative variables) between control group and intervention to check that there are no significant differences between groups.

Finally, the investigators will compare the outcome variables (outcomes) between groups using the chi-square test and the investigators will also do a multivariate analysis (Cox regression) introducing in the model adjustment variables: socio-demographic, risk areas and covariates mentioned above, and considering the time to the event of the outcome variables: admission, fall, sore or infection, institutionalization, and success. For the variable quality of life the investigators will compare the scores (averages and percentiles) of the scale between control group and intervention and also at the beginning and end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients included in the primary care home care program

Exclusion Criteria:

* refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modification of the number of visits to hospital centers, emergency consultations, falls, sores and infections of the study participants. | 1 year
  Data will be collected in relation to the number of hospital visits and emergency visits to calculate avoidable visits. Events such as falls, the presence of sores and / or infections of the study participants will be compiled, taking into account their inclusion in the intervention group or control group to which they have been assigned. The data will be extracted from the clinical history (eCAP) according to the corresponding diagnosis.

SECONDARY OUTCOMES:
Rate of admissions and visits to preventable hospital emergencies | 1 year
  Calculation of the rate of preventable hospital admissions and hospital visits in patients included in the ATDOM program. The number of visits to hospital centers and the number of visits to the emergency services as recorded in the medical record (eCAP) will be recorded.
Infections and sores | 1 year
  Frequency of infections and / or sores in patients included in the ATDOM program according to their inclusion in the control or intervention group. The corresponding diagnosis will be taken into account according to the medical record (eCAP).
Quality of live in ATDOM patients | 1 year
  Modification in the quality of life in the patients included in the ATDOM program according to their inclusion in the intervention or control group. Quality of life will be assessed according to the EuroQol-5D index (validated questionnaire)
Sores, falls, hospital admissions, final institutionalization and death. | 1 year
  Register of sores, falls, hospital admissions, institutionalization and registered deaths of the participants according to intervention or control group. The data will be collected according to registration in the clinical history (eCAP) through corresponding diagnoses.
Risk management in ATDOM patients | 1 year
  Changes in risk management in patients with ATDOM through the implementation of safe practices based on the rapid identification and prioritization of critical areas through a visual risk map. For the evaluation of this indicator, the implementation of nursing care plans will be quantified. The implementation of nursing care plans orients towards prevention measures and improving the quality of care. Nursing care plans are a tool available in the medical record (eCAP) from which preventive activities and care based on clinical evidence can be established.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rey-Reñones, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
not yet decided as future studies are being considered and may be considered
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: The data will be entered on the IDIAP J Gol institution platform
URL: https://www.idiapjgol.org/index.php/ca/

REFERENCES:
- [Derived] Hernandez-Vidal N, Pujol-Vidal M, Mengibar-Garcia Y, Ayala-Villuendas D, Contel-Segura JC, Martinez-Torres S, Bordas A, Oriol-Colominas E, Martin-Vergara N, Martin-Lujan F, Astier-Pena MP, Gens-Barbera M. Design, Implementation, and Evaluation of Healthcare Visual Map Tool for Health Workers to Improve Quality of Life of Home Care Patients: Study Protocol. Healthcare (Basel). 2025 Mar 13;13(6):626. doi: 10.3390/healthcare13060626. PMID 40150476